CLINICAL TRIAL: NCT06614686
Title: A Single-arm, Open-label Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of U87 in Patients With Advanced Malignant Head and Neck Tumors
Brief Title: U87 CAR-T in Patients With Advanced Head and Neck Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U87-01
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Nasopharynx Cancer; Head and Neck Cancer
Keywords: Chimeric Antigen Receptor T Cell; U87
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- U87 autologous CAR T-cell injection (Experimental): Two stages: dose escalation and dose expansion
  Interventions: Drug: U87 autologous CAR T-cell

INTERVENTIONS:
Drug: U87 autologous CAR T-cell — Treatment with U87 chimeric antigen receptor T-cell infusion.

SUMMARY:
This is a single-arm, open-label clinical study to evaluate the safety, tolerability, and efficacy of U87 injection solution in patients with advanced malignant head and neck tumors.

DETAILED DESCRIPTION:
Following consent, patients must have tumor tissue evaluated by IHC assay. Patients meeting all eligibility criteria will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of investigational drug product (U87). Following manufacture of the drug product, subjects will receive preconditioning prior to U87 infusion. All subjects will be asked to continue to undergo long-term gene safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects have provided informed consent, understanding the study's risks and benefits, and are willing to complete the study procedures.
2. Age between 18 and 70 years old at the time of consent, inclusive, and open to both genders.
3. ECOG performance status of 0-1.
4. Anticipated survival of at least 12 weeks.
5. Histologically or cytologically confirmed advanced malignant head and neck cancer patients with no effective standard treatments available
6. Positive Trop2 expression (intensity ≥2+, expression rate ≥40%) in tumor tissue samples within 2 years prior to consent or from recent biopsies.
7. At least one measurable tumor lesion according to RECIST 1.1.
8. Suitable venous access for mononuclear cell collection.
9. Adequate major organ function.
10. Negative pregnancy test for women of reproductive age at screening; sexually active subjects must agree to use effective contraception during the study and for one year after the last CAR-T cell infusion.

Exclusion Criteria:

1. Inadequate washout period from prior anti-cancer treatments before leukapheresis.
2. Receipt of live or attenuated vaccines within 4 weeks prior to leukapheresis or planned receipt during the study.
3. Major surgery or significant trauma within 4 weeks prior to leukapheresis or planned during the study.
4. Previous Trop2-targeted CAR-T/TCR-T cell therapy or other cellular treatments, or therapeutic cancer vaccines.
5. Symptomatic brain metastases or leptomeningeal metastases deemed ineligible by the investigator.
6. Active infection requiring intravenous anti-infective therapy.
7. Positive for HBsAg, HBeAg, HBV-DNA, HCV-Ab, HCV-RNA, TP-Ab, HIV antibodies, or elevated EBV-DNA, CMV-DNA.
8. Primary immunodeficiency or active autoimmune disease.
9. Chronic use of systemic corticosteroids or immunosuppressants within 7 days before leukapheresis, except for local, ophthalmic, intra-articular, intranasal, or inhaled treatments.
10. Prior treatment-related adverse effects not recovered to CTCAE v5.0 grade ≤1 or specified levels, except for non-safety risk toxicities.
11. History of interstitial lung disease, interstitial pneumonia, pulmonary inflammation, or extensive thoracic radiotherapy.
12. Allergy to protein drugs or multiple medications.
13. Other untreated malignancies within 5 years prior to study drug use. History of immune deficiency, hematopoietic stem cell/organ transplantation. Uncontrollable third-space fluid accumulation.
14. Severe cardiovascular or cerebrovascular disease history, including NYHA class ≥II heart failure, uncontrolled hypertension, or recent severe events.

    Pregnant or breastfeeding women.
15. Uncontrollable psychiatric history.
16. Other conditions deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after U87 CAR-T cells infusion [Safety and Tolerability] | 28 days post administration of CAR-T-cells
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

SECONDARY OUTCOMES:
Pharmacokinetics of U87 CAR-T cells | 2 years post CAR T cell infusion
  Time at the maximal concentration(Tmax)
Pharmacokinetics of U87 CAR-T cells | 2 years post CAR T cell infusion
  Area under the concentration-time curve(AUC)
Pharmacokinetics of U87 CAR-T cells | 2 years post CAR T cell infusion
  The maximal concentration of eripheral blood (Cmax)
Pharmacodynamics of U87 CAR-T cells | 2 years post CAR T cell infusion
  Concentration levels of CAR-T-related serum cytokines such as IL-6, IFN γ, ferritin and CRP at each time point
Objective Response Rate (ORR), as assessed by Investigators | 2 years post CAR T cell infusion
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Duration of response (DOR), as assessed by Investigators | 2 years post CAR T cell infusion
  Duration of response (DOR) is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Overall survival (OS) | 2 years post CAR T cell infusion
  Overall Survival (OS) was defined as the time from the date of first infusion of U87 to the date of death due to any cause.
Progression-free survival (PFS), as assessed by Investigators | 2 years post CAR T cell infusion
  Progression-free survival (PFS) was defined as the time from the date of randomization to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.
Disease control rate (DCR), as assessed by Investigators | 2 years post CAR T cell infusion
  Disease control rate (DCR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye ENT Hospital of Fudan University, Shanghai, China